CLINICAL TRIAL: NCT06232642
Title: The Effects of Lactoferrin and Iron-enriched Whey on Iron Status of Active Collegiate Females
Brief Title: Effects of Lactoferrin-enriched Whey on Iron Status in Females
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Collaborators: Glanbia Nutritionals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13314
Record Dates: First submitted 2024-01-04; First posted 2024-01-31 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-04

CONDITIONS: Serum Ferritin
Keywords: Lactoferrin; Iron; Serum Ferritin; Iron Status
MeSH Terms: interventions — Lactoferrin; Iron; Vitamin B 12; Whey Proteins

STUDY DESIGN:
Intervention Model Description: The study has three arms to which participants will be randomly assigned to:
  Arm 1: A lactoferrin- (200 mg), iron (6 mg) and Vitamin B12 (5.2µg)- enriched whey drink (10 g protein; FerriUpTM).
  Arm 2: A protein control (rice protein containing drink matched for protein, iron and B12).
  Arm 3: A lactoferrin control (maltodextrin containing drink matched for lactoferrin, iron, and B12).
  The parallel design 16 weeks in length with blood draws before and after intervention period to assess iron status, and markers of iron metabolism and inflammation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Supplement arms will be marked with a random number code assigned by a non-participating researcher immediately after supplements are prepared. Supplements will be provided to participants in unmarked sachets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lactoferrin in Whey Protein (Active Comparator): Lactoferrin (200 mg), iron (6 mg), and B12 (5.2 ug) in a whey protein isolate drink (20 grams of protein) to be taken 2 times daily; once before the morning meal and once before the evening meal.
  Interventions: Dietary Supplement: Lactoferrin, iron and B12 in Whey Protein
- Lactoferrin in Rice Protein (Active Comparator): Lactoferrin (200 mg), iron (6 mg), and B12 (5.2 ug) in a rice protein drink (20 grams of protein) to be taken 2 times daily; once before the morning meal and once before the evening meal.
  Interventions: Dietary Supplement: Lactoferrin, Iron and B12 in Rice Protein
- Lactoferrin Control (Active Comparator): Lactoferrin (200 mg), iron (6 mg), and B12 (5.2 ug) in a maltodextrin drink (0 grams of protein) to be taken 2 times daily; once before the morning meal and once before the evening meal.
  Interventions: Dietary Supplement: Lactoferrin, Iron and B12 in Maltrodextrin

INTERVENTIONS:
Dietary Supplement: Lactoferrin, iron and B12 in Whey Protein — Chocolate Flavored Whey Protein Isolate Powder with (200mg Lactoferrin, 6 mg Iron, 5.2 ug B12)
  Arms: Lactoferrin in Whey Protein
Dietary Supplement: Lactoferrin, Iron and B12 in Rice Protein — Chocolate Flavored Rice Protein Isolate with (200mg Lactoferrin, 6mg Iron, 5.2 ug B12)
  Arms: Lactoferrin in Rice Protein
Dietary Supplement: Lactoferrin, Iron and B12 in Maltrodextrin — Chocolate Flavored (200mg Lactoferrin, 6 mg Iron, 5.2 ug B12)
  Arms: Lactoferrin Control

SUMMARY:
The goal of this work is to study the effects of twice daily ingestion of a whey protein, rice protein, or maltodextrin drink enriched with lactoferrin- (200 mg), iron (6 mg) and vitamin B12 (5.2 µg) for 16-weeks on iron metabolism and inflammatory markers in active young females. It is expected that the females consuming containing lactoferrin-, iron, and vitamin B12-enriched whey will 1) improve serum ferritin status; 2) reduce inflammation; 3) improve markers of iron metabolism, such as Hemoglobin (Hb), red blood cell count (RBC) and hematocrit (Hc) compared to women who consume the rice protein or maltodextrin control drink. Blood will be drawn before the beginning of the supplemental period (week 0) and end the end of the intervention phase (week 16).

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE

Iron deficiency is a major cause of disease burden worldwide, affecting 1-2 billion people globally. While often considered an issue in developing nations, low iron intake is a growing problem in the US and other industrialized nations, particularly affecting women of reproductive age. In the US, 20% of women aged 18-45 have insufficient iron intake (below the EAR of 18 mg/day) and this number that has been growing over the last decades. This is, in part, due to reduced concentrations in foods and lower intakes of iron-containing foods. Moreover, iron-rich food sources also contain vitamin B12, which is an important co-factor in iron metabolism.

There is, therefore, a strong need to develop strategies that can improve iron status in women of reproductive age, given the generally low intakes of iron-containing sources in this demographic. Besides increasing iron intake, a promising strategy to improve iron status is to ingest compounds that can promote iron uptake. A particularly promising compound to increase iron uptake is lactoferrin.

Lactoferrin (LF) is an iron-binding glycoprotein enriched in mammalian milk. LF binds iron with exceptionally high affinity and is transferred via a variety of receptors into and between cells, serum, bile, and cerebrospinal fluid. It also has important immunological properties, particularly being anti-inflammatory and anti-viral.

LF supplementation has shown initial promise for enhancing iron status in women of reproductive age. A previous study on female long-distance runners, a group at heightened risk for iron-deficiency anemia, found that the combined supplementation of lactoferrin and iron was able to maintain serum ferritin (an indicator of iron status) and red blood cell counts, whereas supplementation with iron alone did not maintain serum ferritin levels and red blood cell counts during the 8-week training period.

To ensure proper absorption, LF is best ingested in a dairy matrix. That is because of the presence of an LF receptor in the human small intestine that can bind bovine LF, likely preventing the use of iron by gut pathogens. This, in turn, results in enhanced systemic availability of iron where it can exert beneficial tissue effects and contribute to adequate iron status.

There is also evidence from in vitro work to suggest that lactoferrin can have anti-inflammatory properties, which could further improve serum iron and hemoglobin concentrations as inflammation negatively impacts iron metabolism. However, more clinical nutrition work is certainly needed to study these potential beneficial effects of LF.

2. STUDY OBJECTIVES

1. To determine the effects of lactoferrin & iron supplementation in whey protein matrix on markers of iron absorption (serum ferritin) compared to a lactoferrin, iron, vitamin b12 and non-milk protein control (rice protein) and a lactoferrin, iron, vitamin b12 control without protein (maltodextrin).
2. To determine the effects of lactoferrin & iron supplementation in whey protein matrix on markers of iron metabolism (RBC, Hb, Hc) compared to a lactoferrin, iron, vitamin b12 and non-milk protein control (rice protein) and a lactoferrin, iron, vitamin b12 control without protein (maltodextrin).
3. To determine the effects of lactoferrin & iron supplementation in whey protein matrix on plasma inflammatory markers (IL-6, TNF-α, and C-reactive protein) compared to a lactoferrin, iron, vitamin b12 and non-milk protein control (rice protein) and a lactoferrin, iron, vitamin b12 control without protein (maltodextrin).

3. DESIGN AND PROCEDURES

3.1 Study duration Participant involvement will be 17 weeks. Week one, participants will go through the initial screening process. participants will consume two servings of supplement per day for the remaining 16 weeks.

3.2 Participants We will recruit 90 physically active female participants between 18-30 yrs, who are physically active (>2 days/week) with a BMI ≥18 and ≤30 kg/m2.

3.3 Description of study visits

Pre-screening (week 1. 15 minutes): Interested participants will have access to the informed consent via a link to recruitment materials. Participants that reach out via email or phone will be provided with a REDCap survey link to the screening questions that asks them further details about their health, diet, and sleep (see inclusion/exclusion criteria). Only minimum personal health information will be collected to determine eligibility. Responses will be reviewed by a study team member (all study team members will have completed the necessary CITI training) and potentially eligible candidates will be contacted to schedule a consent/screening visit. The pre-screen is to confirm that the participant meets most of the criteria before the subject is scheduled for a consent meeting. This will limit subject and research staff time burden. Information gathered will not be attached to identifiers and will be deleted if they decide to not participate or do not meet criteria. If participants screen as a "maybe", they will be contacted by phone or email with follow up questions to determine eligibility. Participants who are taking some medications that may interfere, but who are willing to stop cease usage will require a doctor's release to stop taking prescription medications.

Consent (Week 1. Duration: 1 hour): This visit will take place at the Center for Human Nutrition Studies or will happen virtually (via a tele-call platform such as Zoom). This visit will include the following. Participants will review the consent document with a member of the study team; once all questions have been satisfactorily answered, participants will be asked to sign and date the consent form if participants wish to participate in the study. Participants will be asked to sign the consent form electronically through REDCap using a unique link that is provided to them.

When deemed eligible and contacted, participants can combine the consent visit with the screening visit described below. If participants wish to do so, participants will be asked to come to the Center for Human Nutrition Studies in the morning after an overnight fast, requiring them not to eat or chew gum (nothing but water) 12 hours prior to their arrival. This information will not apply if the investigators do a virtual consent visit first. If participants agree to participate, they will come for the in-person screening visit.

Initial Screening Visit (Week 1. Duration: 1 hour): Assuming participants pre-qualify for the study, and are interested in participating, they will undergo an in-person screening visit. This visit will take place at the Center for Human Nutrition Studies. This visit will be performed in the morning, will last approximately 1 hour, and requires participants not to eat anything or chew gum (nothing but water) for 12 hours prior to their arrival time. This visit will include the following:

* Body mass and height: The investigators will measure their height and body weight to determine their body mass index.
* Blood draw: Participants will have blood drawn from a forearm or hand vein for routine lab analyses (basic metabolic panel and lipid panel), hemoglobinA1c and serum ferritin. The amount drawn will be 15 mL (1 tablespoon) total. If they are of childbearing potential, a pregnancy test will be performed as part of this screening blood draw. It must be negative to participate in this study.
* Questionnaires: If participants agree to participate, participants will be emailed a link with questionnaires to fill out. These questionnaires will ask detailed questions about their diet (7-day food log), potential GI responses such as abdominal discomfort, diarrhea, constipation, gas and bloating using The Gastrointestinal Symptom Rating Scale (GSRS), sleep such as duration and quality, and physical activity patterns, which are part of the screening and/or study process.
* Blood pressure: A blood pressure measurement will be taken using an automated upper arm blood pressure monitor. A total of three measurements will be taken.

Intervention Assignment and Intervention (Week 2 - 17. Duration: 10 min per week): If participants meet the inclusion criteria, participants will be randomly assigned to one of three groups for the duration of the study. The group assignment is random (like the flip of a coin) and participants will not know which group participants are in.

* Lactoferrin in whey group: If participants have been randomly assigned to the lactoferrin in whey protein group, participants they will receive weekly allotments of whey protein concentrate enriched with lactoferrin (a protein found in milk; 200 mg/serving), vitamin B12 (5.2µg/serving) and iron (6 mg/serving). This supplement will come in a flavored powder packaged individually in sachets.
* Lactoferrin alone group: If participants have been randomly assigned to the lactoferrin alone group, they will receive weekly allotments of maltodextrin enriched with B12 (5.2µg/serving), lactoferrin (200mg/serving) and iron (6 mg/serving). This supplement will come in the form of a flavored powder and each serving will be packaged individually in sachets.
* Rice protein group: If participants have been randomly assigned to the whey protein group, they will receive weekly allotments of rice protein concentrate enriched with B12 (5.2µg/serving) and iron (6 mg/serving). This supplement will come in the form of a flavored powder and each serving will be packaged individually in sachets.
* Supplementation schedule: Participants will be asked to take their assigned supplement twice daily, once 30 min before their morning meal, and once between lunch and dinner.
* Weekly pickup: Participants will be asked to pick up the assigned protein supplements at the Center for Human Nutrition Studies once weekly and return the used sachets for record keeping at this visit. They will also be asked to complete questionnaires once weekly regarding GI responses, sleep, and physical activity patterns.
* Tracking: Participants will be asked to mark the time and date that participants take their assigned supplements in an online database called REDcap (described below) so that the research team can determine compliance and provide reminders if necessary.

Mid intervention check-in (Week 9. Duration: 1 hour):

• Questionnaires: 7-day food log The questionnaire will include a 7-day recall of food consumed over the last week including what foods, how much and at about what time.

Final visit (Week 17. Duration: 1 hour): This visit will take place at the Center for Human Nutrition Studies. This visit will be performed in the morning, will last approximately 1 hour, and requires participants not to eat anything or chew gum (nothing but water) for 12 hours prior to their arrival time. This visit will include the following:

* Body mass and height: The investigators will measure their height and body weight to determine their body mass index.
* Blood draw: Participants will have blood drawn from a forearm or hand vein for routine lab analyses and iron status. The amount drawn will be 30 mL (2 tablespoon) total.
* Questionnaires: These questionnaires will ask detailed questions about their diet (7-day food log), GI responses, sleep, and physical activity patterns.
* Blood pressure: A blood pressure measurement will be taken using an automated upper arm blood pressure monitor. A total of three measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex: Female
* Age ≥18 and ≤30 years;
* BMI ≥18 and ≤30 kg/m2;
* For the safety of the participant and proper consent of the procedures, subjects
* must be able to speak and understand English to participate in this study,
* which will be determined at the discretion of study staff;
* Actively engaged in exercise/training ≥3 and ≤12 times per week with each session being from ≥30min to ≤3 hours in length of moderate to vigorous activity. activities that meet this criterion may include but are not limited to: hiking, weightlifting, volleyball, basketball, soccer, or others sport or activities' that involves strenuous physical activity

Exclusion Criteria:

* Use of medications or supplements that are known to affect the study outcome measures (e.g., NSAIDs, corticosteroids, iron containing supplements) or increase the risk of study procedures (e.g., anticoagulants) that cannot be temporarily discontinued for this study.
* Allergy to rice and/or whey protein.
* Pregnant or lactating.
* >7 meals/week containing red meat and/or shellfish (iron-rich foods).
* Hb1Ac >6.4%
* Consuming >14 alcoholic drinks per week;
* Use of cigarettes (or other tobacco products) in last 3 months;
* Diagnoses of active malignancy, congestive heart failure, diabetes mellitus or chronic obstructive pulmonary disease;
* Any inflammatory diseases (e.g., autoimmune diseases, coeliac disease, glomerulonephritis, hepatitis, inflammatory bowel disease, arthritis).
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Serum Ferritin | Tested at week 0 before supplementation begins, and week 16 after the final supplements have been taken.
  Free Serum Ferritin measured via enzymatic detection at LabCorp Inc. as proxy of iron absorption.

SECONDARY OUTCOMES:
Inflammatory cytokine biomarker (IL-6) concentrations in plasma samples | Tested at week 0 before supplementation begins, and week 16 after the final supplements have been taken.
  Plasma Inflammatory Biomarker, measured via multiplex electro-chemiluminescence at Utah State University.
Inflammatory cytokine biomarker (C-reactive protein) concentrations in plasma samples | Tested at week 0 before supplementation begins, and week 16 after the final supplements have been taken.
  Plasma Inflammatory Biomarker, measured via multiplex electro-chemiluminescence at Utah State University.
Inflammatory cytokine biomarker (TNF-alpha) concentrations in plasma samples | Tested at week 0 before supplementation begins, and week 16 after the final supplements have been taken.
  Plasma Inflammatory Biomarker, measured via multiplex electro-chemiluminescence at Utah State University.
Marker of Iron metabolism Red Blood Cell Count | Tested at week 0 before supplementation begins, and on week 16 after the final supplements have been taken.
  Marker of Iron Metabolism determined via Metabolomics analysis via LC/tandem MS (LC-MS/MS; Sciex QTRAP 7500). Metabolites will be identified by automated comparison of the ion features in the experimental samples to a reference library of chemical standards that include retention time, molecular weight (m/z), preferred adducts, and in-source fragments as well as associated MS spectra.
Marker of Iron metabolism Hematocrit | Tested at week 0 before supplementation begins, and week 16 after the final supplements have been taken.
  Marker of Iron Metabolism determined via Metabolomics analysis via LC/tandem MS (LC-MS/MS; Sciex QTRAP 7500). Metabolites will be identified by automated comparison of the ion features in the experimental samples to a reference library of chemical standards that include retention time, molecular weight (m/z), preferred adducts, and in-source fragments as well as associated MS spectra.
Marker of Iron metabolism Hemoglobin | Tested on week 1 before supplementation begins, and week 16 after the final supplements have been taken.
  Marker of Iron Metabolism determined via Metabolomics analysis via LC/tandem MS (LC-MS/MS; Sciex QTRAP 7500). Metabolites will be identified by automated comparison of the ion features in the experimental samples to a reference library of chemical standards that include retention time, molecular weight (m/z), preferred adducts, and in-source fragments as well as associated MS spectra.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Any de-identified collected data through RedCap and wet-lab assays will be made available upon publication.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: From January 2025, and indefinitely afterward.
Access Criteria: Freely Available

REFERENCES:
- [Background] Sun H, Weaver CM. Decreased Iron Intake Parallels Rising Iron Deficiency Anemia and Related Mortality Rates in the US Population. J Nutr. 2021 Jul 1;151(7):1947-1955. doi: 10.1093/jn/nxab064. PMID 33834234
- [Background] Rosa L, Lepanto MS, Cutone A, Siciliano RA, Paesano R, Costi R, Musci G, Valenti P. Influence of oral administration mode on the efficacy of commercial bovine Lactoferrin against iron and inflammatory homeostasis disorders. Biometals. 2020 Jun;33(2-3):159-168. doi: 10.1007/s10534-020-00236-2. Epub 2020 Apr 9. PMID 32274616
- [Background] Rezk M, Dawood R, Abo-Elnasr M, Al Halaby A, Marawan H. Lactoferrin versus ferrous sulphate for the treatment of iron deficiency anemia during pregnancy: a randomized clinical trial. J Matern Fetal Neonatal Med. 2016;29(9):1387-90. doi: 10.3109/14767058.2015.1049149. Epub 2015 Jun 3. PMID 26037728
- [Background] Paesano R, Torcia F, Berlutti F, Pacifici E, Ebano V, Moscarini M, Valenti P. Oral administration of lactoferrin increases hemoglobin and total serum iron in pregnant women. Biochem Cell Biol. 2006 Jun;84(3):377-80. doi: 10.1139/o06-040. PMID 16936810
- [Background] Paesano R, Berlutti F, Pietropaoli M, Goolsbee W, Pacifici E, Valenti P. Lactoferrin efficacy versus ferrous sulfate in curing iron disorders in pregnant and non-pregnant women. Int J Immunopathol Pharmacol. 2010 Apr-Jun;23(2):577-87. doi: 10.1177/039463201002300220. PMID 20646353
- [Background] Omar OM, Assem H, Ahmed D, Abd Elmaksoud MS. Lactoferrin versus iron hydroxide polymaltose complex for the treatment of iron deficiency anemia in children with cerebral palsy: a randomized controlled trial. Eur J Pediatr. 2021 Aug;180(8):2609-2618. doi: 10.1007/s00431-021-04125-9. Epub 2021 May 28. PMID 34101010
- [Background] Mikulic N, Uyoga MA, Mwasi E, Stoffel NU, Zeder C, Karanja S, Zimmermann MB. Iron Absorption is Greater from Apo-Lactoferrin and is Similar Between Holo-Lactoferrin and Ferrous Sulfate: Stable Iron Isotope Studies in Kenyan Infants. J Nutr. 2020 Dec 10;150(12):3200-3207. doi: 10.1093/jn/nxaa226. PMID 32886113
- [Background] Lonnerdal B, Du X, Jiang R. Biological activities of commercial bovine lactoferrin sources. Biochem Cell Biol. 2021 Feb;99(1):35-46. doi: 10.1139/bcb-2020-0182. Epub 2020 Jul 24. PMID 32706983
- [Background] Lepanto MS, Rosa L, Cutone A, Conte MP, Paesano R, Valenti P. Efficacy of Lactoferrin Oral Administration in the Treatment of Anemia and Anemia of Inflammation in Pregnant and Non-pregnant Women: An Interventional Study. Front Immunol. 2018 Sep 21;9:2123. doi: 10.3389/fimmu.2018.02123. eCollection 2018. PMID 30298070
- [Background] Kruzel ML, Actor JK, Boldogh I, Zimecki M. Lactoferrin in health and disease. Postepy Hig Med Dosw (Online). 2007;61:261-7. PMID 17507874
- [Background] Ke C, Lan Z, Hua L, Ying Z, Humina X, Jia S, Weizheng T, Ping Y, Lingying C, Meng M. Iron metabolism in infants: influence of bovine lactoferrin from iron-fortified formula. Nutrition. 2015 Feb;31(2):304-9. doi: 10.1016/j.nut.2014.07.006. Epub 2014 Aug 1. PMID 25592008
- [Background] El-Hawy MA, Abd Al-Salam SA, Bahbah WA. Comparing oral iron bisglycinate chelate, lactoferrin, lactoferrin with iron and iron polymaltose complex in the treatment of children with iron deficiency anemia. Clin Nutr ESPEN. 2021 Dec;46:367-371. doi: 10.1016/j.clnesp.2021.08.040. Epub 2021 Sep 29. PMID 34857222
- [Background] El Amrousy D, El-Afify D, Elsawy A, Elsheikh M, Donia A, Nassar M. Lactoferrin for iron-deficiency anemia in children with inflammatory bowel disease: a clinical trial. Pediatr Res. 2022 Sep;92(3):762-766. doi: 10.1038/s41390-022-02136-2. Epub 2022 Jun 9. PMID 35681097
- [Background] Artym J, Zimecki M, Kruzel ML. Lactoferrin for Prevention and Treatment of Anemia and Inflammation in Pregnant Women: A Comprehensive Review. Biomedicines. 2021 Jul 27;9(8):898. doi: 10.3390/biomedicines9080898. PMID 34440102
- [Background] Pasricha SR, Tye-Din J, Muckenthaler MU, Swinkels DW. Iron deficiency. Lancet. 2021 Jan 16;397(10270):233-248. doi: 10.1016/S0140-6736(20)32594-0. Epub 2020 Dec 4. PMID 33285139
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Miller EM. Iron status and reproduction in US women: National Health and Nutrition Examination Survey, 1999-2006. PLoS One. 2014 Nov 6;9(11):e112216. doi: 10.1371/journal.pone.0112216. eCollection 2014. PMID 25375360
- [Background] Koury MJ, Ponka P. New insights into erythropoiesis: the roles of folate, vitamin B12, and iron. Annu Rev Nutr. 2004;24:105-31. doi: 10.1146/annurev.nutr.24.012003.132306. PMID 15189115
- [Background] Koikawa N, Nagaoka I, Yamaguchi M, Hamano H, Yamauchi K, Sawaki K. Preventive effect of lactoferrin intake on anemia in female long distance runners. Biosci Biotechnol Biochem. 2008 Apr;72(4):931-5. doi: 10.1271/bbb.70383. Epub 2008 Apr 7. PMID 18391460
- [Background] Suzuki YA, Shin K, Lonnerdal B. Molecular cloning and functional expression of a human intestinal lactoferrin receptor. Biochemistry. 2001 Dec 25;40(51):15771-9. doi: 10.1021/bi0155899. PMID 11747454
- [Background] Shin K, Wakabayashi H, Yamauchi K, Yaeshima T, Iwatsuki K. Recombinant human intelectin binds bovine lactoferrin and its peptides. Biol Pharm Bull. 2008 Aug;31(8):1605-8. doi: 10.1248/bpb.31.1605. PMID 18670097
- [Background] Berlutti F, Schippa S, Morea C, Sarli S, Perfetto B, Donnarumma G, Valenti P. Lactoferrin downregulates pro-inflammatory cytokines upexpressed in intestinal epithelial cells infected with invasive or noninvasive Escherichia coli strains. Biochem Cell Biol. 2006 Jun;84(3):351-7. doi: 10.1139/o06-039. PMID 16936806
- [Background] Griffin IJ. The Effects of Different Forms of Lactoferrin on Iron Absorption. J Nutr. 2020 Dec 10;150(12):3053-3054. doi: 10.1093/jn/nxaa314. No abstract available. PMID 33188407
- [Background] Kell DB, Heyden EL, Pretorius E. The Biology of Lactoferrin, an Iron-Binding Protein That Can Help Defend Against Viruses and Bacteria. Front Immunol. 2020 May 28;11:1221. doi: 10.3389/fimmu.2020.01221. eCollection 2020. PMID 32574271